CLINICAL TRIAL: NCT00532220
Title: Study Into the Effect of Ibandronate for the Treatment of Bone Marrow Edema in Relation to Spontaneous or Non-traumatic Osteonecrosis of the Knee: A Randomized Double-blind, Placebo-controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Christian Meier, PD, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ro 200-5450
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Osteonecrosis of the Knee; Bone Marrow Edema of the Knee
Keywords: osteonecrosis; bone marrow edema; ibandronate; bisphosphonate; knee
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Ibandronate IV
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibandronate IV — Ibandronate IV (Bonviva® IV), 10.5 mg divided in 4 single infusions within 2 weeks(1x1.5 mg, 3x3 mg), followed by a fifth infusion after 3 months (V4)
  Arms: A
Drug: Placebo — Placebo IV, divided in 4 single infusions within 2 weeks, followed by a fifth infusion after 3 months (V4)
  Arms: B

SUMMARY:
BACKGROUND: Bone marrow edema (BME) in the knee occurs as a localized inflammatory disease in relation to spontaneous or non-traumatic osteonecrosis (ON). Prognosis of BME/ON in the course after knee arthroscopy appears to be poor and in most cases results in knee arthroplasty. Treatment options of ON depend in general on the size of the lesion. Smaller lesions are managed by mechanical unloading and use of non-steroidal anti-inflammatory drugs, larger lesion in general requires osteotomy or arthroplasty. In animal studies it has been shown that bisphosphonates prevent resorption of necrotic bone during ischemic necrosis and revascularization. In humans, bisphosphonate treatment has been used successfully in bone marrow oedema and avascular necrosis of the femoral head.

In an observational study using bisphosphonates (ibandronate, pamidronate) in patients with either spontaneous or (believed to be) arthroscopy-induced BME of the knee a significant rapid and sustained pain relief was observed with a mean decrease on the pain scale on the visual analogue scale of over 60% after 3 months and of 80% after 6 months. Our experience suggests an apparent beneficial effect of amino-bisphosphonates in the treatment of BME of the knee.

AIM: This randomized, double-blind, placebo-controlled study aims to provide data on clinical, biochemical and radiological outcome of patients with bone marrow edema in relation to spontaneous or arthroscopy-induced ON of the knee treated with ibandronate or placebo.

ENDPOINTS: The primary objective is to demonstrate the superiority of treatment with ibandronate compared to placebo regarding clinical outcome (pain [VAS score]) in spontaneous or arthroscopy-induced BME/ON of the knee after 12 weeks. Secondary objectives include a) clinical outcome (pain [VAS score]) after 24 weeks, b) the evaluation of the radiological outcome (MRI scan) at 12 and 48 weeks, c) the changes in biochemical markers of bone turnover, and d) the number of salvage therapies needed in case persistence is observed during placebo therapy.

METHODS: The study is designed as a single-center, randomized double-blind, placebo-controlled trial. A total number of 30 patients with BME/ON will be recruited. Each patient will be randomized in a 1:1 ratio to receive ibandronate IV or placebo IV. Additionally, all patients will receive 500 mg calcium and 400 IU vitamin D per day throughout the study, and diclofenac/esomeprazole for initial 3 months (blinded treatment duration 24 weeks). Baseline and follow-up data collection will contain all variables needed for evaluation of clinical, biochemical and radiological evaluation of treatment efficacy.

EXPECTED RESULTS: We hypothesize that treating patients with BME/ON of the knee, therapy with ibandronate will be superior in reducing pain, and radiological findings as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with newly diagnosed BME in relation to ON, confirmed by MRI scan

Exclusion Criteria:

* Baseline renal insufficiency (calculated creatinine clearance <50 ml/min)
* Baseline hypocalcemia (serum calcium <2.0 mmol/l)
* Premenopausal women without adequate contraception
* Hypersensitivity to bisphosphonates
* Prior treatment with bisphosphonates within the last 2 years prior to randomization
* Prior treatment with calcitonin within the last month prior to randomization
* Treatment with any investigational drug within 30 days prior to randomization
* Any medical or psychiatric condition which, in the opinion of the investigator, would preclude the participant from adhering to the protocol or completing the trial per protocol
* Unable to provide informed consent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
clinical outcome (pain [VAS score]) | 12 weeks

SECONDARY OUTCOMES:
clinical outcome (pain [VAS score]) | 24 weeks
radiological outcome (MRI knee) | 12 and 24 weeks
number of salvage therapies needed in case persistence is observed during placebo therapy | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meier, MD, Principal Investigator — University Hospital, Basel, Switzerland; Marius E Kraenzlin, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland